CLINICAL TRIAL: NCT00589121
Title: A Phase II Trial of Image Guided Preoperative Radiotherapy for Primary Soft Tissue Sarcomas of the Extremity
Brief Title: Image-Guided Radiation Therapy in Treating Patients With Primary Soft Tissue Sarcoma of the Shoulder, Arm, Hip, or Leg
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0630; CDR0000582196
Record Dates: First submitted 2008-01-05; First posted 2008-01-09 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2018-06

CONDITIONS: Lymphedema; Musculoskeletal Complications; Radiation Fibrosis; Radiation Toxicity; Sarcoma
Keywords: radiation fibrosis; radiation toxicity; lymphedema; musculoskeletal complications; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; adult extraskeletal chondrosarcoma; stage III adult soft tissue sarcoma
MeSH Terms: conditions — Lymphedema; Radiation Fibrosis Syndrome; Radiation Injuries; Sarcoma; Chondrosarcoma, Extraskeletal Myxoid | interventions — Drug Therapy; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A - Chemotherapy (Experimental): Radiation therapy with neoadjuvant or adjuvant or concurrent or interdigitated chemotherapy followed by surgery followed by, for patients with positive margins, radiation therapy boost
  Interventions: Drug: Chemotherapy; Radiation: Radiation therapy; Procedure: Surgery
- Cohort B - No Chemotherapy (Experimental): Radiation therapy followed by surgery followed by, for patients with positive margins, radiation therapy boost
  Interventions: Radiation: Radiation therapy; Procedure: Surgery

INTERVENTIONS:
Drug: Chemotherapy — Up to 6 courses of investigator's choice of neoadjuvant, adjuvant, concurrent, or interdigitated chemotherapy
  Arms: Cohort A - Chemotherapy
Radiation: Radiation therapy — Preoperative IGRT (3D-CRT or IMRT): If receiving neoadjuvant or adjuvant chemotherapy or no chemotherapy: 50 Gy (2 Gy once a day, 5 times a week). If receiving concurrent or interdigitated chemotherapy: 44 Gy (2 Gy once a day, 5 times a week). Postoperative radiotherapy boost for patients with positive margins following surgery: 16 Gy (2 Gy once a day, 5 times a week) external beam radiation therapy or 16 Gy at ≤ 80 cGy per hour brachytherapy or 3.4 Gy/fraction in 4 fractions brachytherapy or 10-12.5 Gy in a single fraction intraoperative radiation therapy boost.
Procedure: Surgery — Resection of the sarcoma with the goal of having negative pathologic margins. Every effort should be made to have limb preservation surgery unless there is documented evidence of tumor progression that would require amputation for an appropriate negative margin resection. All lesions of the extremities should be treated with wide excision.

SUMMARY:
RATIONALE: Image-guided radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a lower dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase II trial is studying the side effects and how well image-guided radiation therapy works in treating patients with primary soft tissue sarcoma of the shoulder, arm, hip, or leg.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the effect of reduced radiation volume using image-guided radiotherapy (IGRT) on lymphedema ≥ grade 2, subcutaneous fibrosis, and joint stiffness at 2 years in patients with primary soft tissue sarcoma of the extremity.

Secondary

* To estimate the rates of other grade 3-5 adverse events as measured by Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0.
* To determine the pattern of first failure, including local failure (in-field, marginal, and outside-field failure), regional failure, distant failure, and death without disease progression.
* To estimate the rates of local failure, local-regional failure, distant failure, distant disease-free survival, disease-free survival, overall survival, and second primary tumor.
* To estimate the rate of wound complications.
* To correlate the degree of late radiation morbidity (defined as any lymphedema, subcutaneous fibrosis, or joint stiffness) at 2 years with scores on the clinical measure, Musculoskeletal Tumor Rating Scale (MSTS).

OUTLINE: This is a multicenter study.

* Neoadjuvant radiotherapy: Patients are assigned to 1 of 2 treatment groups (group 1 closed to accrual as of 01/08/10).

  * Group 1 (closed to accrual as of 01/08/10): Patients undergo 3-D conformal radiotherapy (3D-CRT) or intensity-modulated therapy (IMRT) once daily, 5 days a week, for 4½-5 weeks. Patients also receive up to 6 courses of neoadjuvant, adjuvant, concurrent, or interdigitated chemotherapy.
  * Group 2: Patients undergo 3D-CRT or IMRT once daily, 5 days a week, for 5 weeks.
* Surgery: At 4-8 weeks after completion of neoadjuvant radiotherapy, patients undergo surgical resection of the tumor. Patients with positive tumor margins (residual tumor) undergo intraoperative radiotherapy boost or proceed to adjuvant radiotherapy within 2 weeks after surgery.
* Adjuvant radiotherapy: Patients undergo either external-beam radiotherapy (EBRT) once daily for 8 fractions or brachytherapy.

After completion of study treatment, patients are followed at least every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary soft tissue sarcoma of the upper extremity (including shoulder) or lower extremity (including hip)

  * Incisional or core biopsy required within the past 8 weeks
* No histopathological diagnosis of any of the following:

  * Rhabdomyosarcoma
  * Extraosseous primitive neuroectodermal tumor (PNET)
  * Soft tissue Ewing sarcoma
  * Osteosarcoma
  * Kaposi sarcoma
  * Angiosarcoma
  * Aggressive fibromatosis (desmoid tumor)
  * Dermatofibrosarcoma protuberans
  * Chondrosarcoma

    * Extraskeletal myxoid chondrosarcoma allowed
* Tumor must be surgically resectable, as determined by a surgeon within the past 8 weeks

  * Limb-preservation surgery alone would not provide adequate local control, as determined by the surgeon
* No sarcoma of the hand, foot, head, neck, or intra-abdominal or retroperitoneal region or body wall
* No sarcoma ≥ 32 cm in any direction
* No lymph node or distant metastases, according to the following within the past 8 weeks:

  * History/physical examination, including a detailed description of the location, size, and stage of the sarcoma
  * MRI with contrast of the primary tumor

    * The maximum dimension of the primary tumor is measured in MRI images
  * CT scan of the chest

    * Multiple pulmonary nodules < 8 mm without a histological diagnosis detected incidentally on a non-screening CT scan may be allowed
  * CT scan with contrast of the abdomen and pelvis in patients with intermediate- or high-grade sarcoma of the upper thigh
* No recurrent tumor after prior potentially curative therapy

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL (transfusion or other intervention allowed)
* Bilirubin ≤ 1.5 mg/dL*
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2 times upper limit of normal*
* Serum creatinine ≤ 1.6 mg/dL OR creatinine clearance ≥ 55 mL/min*
* Left ventricular ejection fraction (LVEF) ≥ 50% by multiple gated acquisition scan (MUGA) or echocardiogram*
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other invasive malignancy within the past 3 years, except nonmelanomatous skin cancer or carcinoma in situ of the breast, oral cavity, or cervix
* No severe, active co-morbidity, including any of the following*:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial infection or fungal infection requiring intravenous antibiotics
  * Acquired Immune Deficiency Syndrome (AIDS) or immunocompromised patients

    * HIV testing not required
* No NCI CTCAE v 3.0 grade 3-4 electrolyte abnormalities, including any of the following*:

  * Calcium < 7 mg/dL or > 12.5 mg/dL
  * Glucose < 40 mg/dL or > 250 mg/dL
  * Magnesium < 0.9 mg/dL or > 3 mg/dL
  * Potassium < 3mmol/L or > 6 mmol/L
  * Sodium < 130 mmol/L or > 155 mmol/L NOTE: *Applies to group 1 only, which was closed to accrual as of 01/08/10)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior excisional biopsy in which the majority of the tumor (≥ 50%) is removed
* No prior radiotherapy to the region of the study cancer that would result in overlap of radiotherapy fields
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dian Wang, MD, PhD, Principal Investigator — Medical College of Wisconsin; Scott Okuno, MD, Study Chair — Mayo Clinic; Burton L. Eisenberg, MD, Study Chair — Norris Cotton Cancer Center; John M. Kane, MD, Study Chair — Roswell Park Cancer Institute; David G. Kirsch, MD, PhD, Study Chair — Duke Cancer Institute
Locations (17):
- United States (14):
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Norton Suburban Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (3):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Wang D, Harris J, Kraybill WG, Eisenberg B, Kirsch DG, Ettinger DS, Kane JM 3rd, Barry PN, Naghavi A, Freeman CR, Chen YL, Hitchcock YJ, Bedi M, Salerno KE, Severin D, Godette KD, Larrier NA, Curran WJ Jr, Torres-Saavedra PA, Lucas DR. Pathologic Complete Response and Clinical Outcomes in Patients With Localized Soft Tissue Sarcoma Treated With Neoadjuvant Chemoradiotherapy or Radiotherapy: The NRG/RTOG 9514 and 0630 Nonrandomized Clinical Trials. JAMA Oncol. 2023 May 1;9(5):646-655. doi: 10.1001/jamaoncol.2023.0042. PMID 36995690
- [Derived] Wang D, Zhang Q, Eisenberg BL, Kane JM, Li XA, Lucas D, Petersen IA, DeLaney TF, Freeman CR, Finkelstein SE, Hitchcock YJ, Bedi M, Singh AK, Dundas G, Kirsch DG. Significant Reduction of Late Toxicities in Patients With Extremity Sarcoma Treated With Image-Guided Radiation Therapy to a Reduced Target Volume: Results of Radiation Therapy Oncology Group RTOG-0630 Trial. J Clin Oncol. 2015 Jul 10;33(20):2231-8. doi: 10.1200/JCO.2014.58.5828. Epub 2015 Feb 9. PMID 25667281

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A - Chemotherapy | Cohort B - No Chemotherapy
Started | 12 | 86
Completed | 10 (Subjects with data available for the analysis are considered to have completed the study.) | 79 (Subjects with data available for the analysis are considered to have completed the study.)
Not Completed | 2 | 7
Not completed — Protocol Violation | 2 | 6
Not completed — No protocol treatment received | 0 | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients who started protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - Chemotherapy | Cohort B - No Chemotherapy | Total
Number analyzed (Participants) | 10 | 79 | 89
Age, Continuous [Median (Full Range); unit: years] | 52 [30 to 71] | 61 [24 to 88] | 61 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 37 | 42
  Male | 5 | 42 | 47

OUTCOME MEASURES:

1. Primary Outcome: Rate of Late Radiation Morbidity (≥ Grade 2 Lymphedema, Subcutaneous Fibrosis, or Joint Stiffness) at 2 Years From the Start of Radiotherapy as Measured by EORTC/RTOG Criteria
Description: The rate of patients with late radiation morbidity (≥ grade 2 lymphedema, subcutaneous fibrosis, or joint stiffness) at 2 years from the start of radiotherapy as measured by EORTC(European Organisation for Research and Treatment of Cancer)/RTOG (Radiation Therapy Oncology Group) criteria. Grade refers to the severity of the morbidity. The RTOG/EORTC Late Radiation Morbidity Scoring Schema assigns Grades 1 through 5 with unique clinical descriptions of severity for each morbidity based on this general guideline: Grade 1 Mild , Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to morbidity.
Time Frame: 2 years after start of treatment (+/- 3 months)
Population: All eligible patients on Cohort B who started study treatment and had an assessment of toxicity at 2 years. (See limitations and caveats, Cohort A is not included.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 57
percentage of participants | 10.5 [2.6 to 18.5]
Statistical Analysis 1: Comparison: Cohort B - No Chemotherapy; Initially designed to test for a 20% absolute improvement from 37% (fixed rate) to 17% using Fisher's exact test, requiring 41 patients per cohort (51 with 20% ineligibility) with 5% type I error and 90% statistical power. During accrual, the sample size for cohort B was increased to 66 (83 with 20% ineligibility) to test for a 15% improvement with 5% type I error and 85% power; Test type: Superiority or Other — The fixed rate of 37% comes from the published National Cancer Institute of Canada trial SR2 (CAN-NCIC-SR2: Phase III Randomized Study of Pre- vs Postoperative Radiotherapy in Curable Extremity Soft Tissue Sarcoma) receiving preoperative radiation therapy without image-guided radiation therapy (IGRT); p = 0.0005, Fisher Exact

2. Secondary Outcome: Local Failure Rate at Two Years
Description: Local failure is defined as the time from registration to date of failure (local progression) or death or last follow-up. Two year rate and 95% confidence interval were estimated by the cumulative incidence method.
Time Frame: From registration to date of failure (local progression) or death or last follow-up. Report at time of primary outcome measure analysis.
Population: All eligible patients on Cohort B who started study treatment. (See limitations and caveats, Cohort A is not included.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 79
percentage of participants | 11.4 [5.6 to 19.6]

3. Secondary Outcome: Regional Failure Rate at Two Years
Description: Regional failure is defined as the time from registration to date of failure (regional progression) or death or last follow-up. Two year rate and 95% confidence interval were estimated by the cumulative incidence method.
Time Frame: From registration to date of failure (regional progression) or death or last follow-up. Report at time of primary outcome measure analysis.
Population: All eligible patients on Cohort B who started study treatment. (See limitations and caveats, Cohort A is not included.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 79
percentage of participants | 0 [0 to 0]

4. Secondary Outcome: Distant Failure Rate at Two Years
Description: Distant failure is defined as the time from registration to date of failure (distant progression) or death or last follow-up. Two year rate and 95% confidence interval were estimated by the cumulative incidence method.
Time Frame: From registration to date of failure (distant progression) or death or last follow-up. Report at time of primary outcome measure analysis.
Population: All eligible patients on Cohort B who started study treatment. (See limitations and caveats, Cohort A is not included.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 79
percentage of participants | 37.3 [26.6 to 48]

5. Secondary Outcome: Distant Disease-free Survival Rate at Two Years
Description: Distant disease-free survival is defined as the time from registration to date of failure (distant progression or death) or last follow-up. Two year rate and 95% confidence interval were estimated by the Kaplan-Meier method.
Time Frame: From registration to date of failure (distant progression or death) or last follow-up. Report at time of primary outcome measure analysis.
Population: All eligible patients on Cohort B who started study treatment. (See limitations and caveats, Cohort A is not included.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 79
percentage of participants | 61.4 [50.6 to 72.2]

6. Secondary Outcome: Disease-free Survival Rate at Two Years
Description: Disease-free survival is defined as the time from registration to date of failure (local, regional, or distant progression or death) or last follow-up. Two year rate and 95% confidence interval were estimated by the Kaplan-Meier method.
Time Frame: From registration to date of failure (local, regional or distant progression or death) or last follow-up. Report at time of primary outcome measure analysis.
Population: All eligible patients on Cohort B who started study treatment. (See limitations and caveats, Cohort A is not included.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 79
percentage of participants | 58.1 [47.1 to 69.0]

7. Secondary Outcome: Overall Survival Rate at Two Years
Description: Overall survival is defined as the time from registration to date of death or last follow-up. Two year survival rate and 95% confidence interval were estimated by the Kaplan-Meier method.
Time Frame: From registration to date of death or last follow-up. Report at time of primary outcome measure analysis.
Population: All eligible patients on Cohort B who started study treatment. (See limitations and caveats, Cohort A is not included.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 79
percentage of participants | 80.6 [71.8 to 89.4]

8. Secondary Outcome: Second Primary Tumor Rate at Two Years
Description: Second primary tumor is defined as the time from registration to date of failure (second primary tumor) or death or last follow-up. Two year rate and 95% confidence interval were estimated by the cumulative incidence method.
Time Frame: From registration to date of failure (second primary tumor) or death or last follow-up. Report at time of primary outcome measure analysis.
Population: All eligible patients on Cohort B who started study treatment. (See limitations and caveats, Cohort A is not included.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 79
percentage of participants | 5.1 [1.7 to 11.7]

9. Secondary Outcome: Late Radiation Morbidity Rate (≥ Grade 2 Lymphedema, Subcutaneous Fibrosis or Joint Stiffness) at 2 Years From the Start of Radiotherapy as Measured by CTCAE v3.0
Description: Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: 2 years after start of treatment (+/- 3 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 57
percentage of participants | 8.8 [1.4 to 16.1]

10. Secondary Outcome: Percentage of Patients With Wound Complications
Description: Estimate rate of patients with acute wound complications with 95% confidence interval assuming binomial distribution.
Time Frame: From date of surgery to 4 months post-surgery
Population: All eligible patients on cohort B that had surgery and a wound assessment. (See limitations and caveats, Cohort A is not included.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 71
percentage of participants | 36.6 [25.4 to 47.8]

11. Secondary Outcome: Pattern of First Failure
Description: Pattern of first failure including local failure (in-field, marginal, and outside-field failure), regional failure, distant failure, and death without disease progression.
Time Frame: From registration to date of local, regional or distant progression. Report at time of primary outcome measure analysis.
Population: All eligible patients on Cohort B who started study treatment. All eligible patients on Cohort B. (See limitations and caveats, Cohort A is not included.)
Measure: Number; unit: participants
Arm/Group | Cohort A - Chemotherapy | Cohort B - No Chemotherapy
Number analyzed (Participants) | 10 | 79
participants
  Local | 1 | 8
  Regional | 0 | 1
  Distant | 1 | 29
  Dead without disease progression | 0 | 2
  Alive without disease progression | 8 | 39

12. Secondary Outcome: Mean Musculoskeletal Tumor Rating Scale (MSTS) by Late Radiation Morbidity at Two Years
Description: The Musculoskeletal Tumor Rating Scale (MSTS) is a measure of physical function across 7 items, completed by the physician (preferably by the Orthopedic Surgeon or Surgical Oncologist) or the physician's designated staff. The 7 items are: pain, range of motion, strength, joint stability, joint deformity, emotional, acceptance, and overall function. Each item is scored from 0-5 (worst possible to best possible condition). The item scores are summed to get the total score which ranges from 0-35.
  Late radiation morbidity is defined as ≥ grade 2 lymphedema, subcutaneous fibrosis, or joint stiffness. Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From start of treatment to 2 years.
Population: All eligible patients on Cohort B who had a 2-year MSTS assessment. (See limitations and caveats, Cohort A is not included.)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Late Radiation Morbitity | Has Late Radiation Toxicity
Number analyzed (Participants) | 18 | 2
units on a scale | 31.3 (4.5) | 25.0 (0)

13. Secondary Outcome: Percentage of Patients With Other CTCAE, v.3.0 Grade 3-5 Adverse Events
Description: as for outcome 9
Time Frame: From start of treatment to last follow-up. Analysis can occur at or after time of primary outcome measure analysis.
Population: All eligible patients on Cohort B who started study treatment. (See limitations and caveats, Cohort A is not included.)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort B - No Chemotherapy
Number analyzed (Participants) | 79
percentage of patients | 38.0 [27.3 to 49.6]

14. Other Pre Specified Outcome: Correlation of Late Radiation Morbidity at 2 Years With the 3 Quality of Life Assessments [Functional Assessment of Cancer Therapy-General (FACTG), Toronto Extremity Salvage Score (TESS), and Sexual Adjustment Questionnaire (SAQ)]
Time Frame: 2 years after start of treatment (+/- 3 months)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Comparison of TESS and the MSTS Scores at 2 Years Between Cohort B Patients and the Preoperative Radiotherapy Patients in the NCIC CTG Trial [National Cancer Institute of Canada Clinical Trials Group]
Time Frame: 2 years after start of treatment (+/- 3 months)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Comparison of SAQ Scores at 2 Years for Cohort A Patients With Cohort B Patients
Time Frame: 2 years after start of treatment (+/- 3 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event (AE) are counted only once for that adverse event. Data is reported for eligible patients with adverse event data who started study treatment.
Arm/Group | Cohort A - Chemotherapy | Cohort B - No Chemotherapy
Serious Adverse Events (participants affected / at risk) | 2/10 | 13/79
Other Adverse Events (participants affected / at risk) | 8/10 | 73/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - Chemotherapy (N=10) | Cohort B - No Chemotherapy (N=79)
Blood disorder (Blood and lymphatic system disorders) | 1 | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Edema limbs (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 0
Infection [other] (Infections and infestations) | 1 | 0
Opportunistic infection (Infections and infestations) | 0 | 1
Skin infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 3
Wound infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1
Arterial injury - Extremity-lower (Injury, poisoning and procedural complications) | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Late RT Toxicity: subcutaneous tissue: NOS (Injury, poisoning and procedural complications) | 0 | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Laboratory test abnormal (Investigations) | 1 | 0
Leukopenia (Investigations) | 1 | 1
Lymphopenia (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 0 | 1
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Late RT Toxicity: joint: NOS (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2
Confusion (Psychiatric disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Vascular disorder (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - Chemotherapy (N=10) | Cohort B - No Chemotherapy (N=79)
Blood disorder (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 | 19
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Premature ventricular contractions (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhea (Gastrointestinal disorders) | 1 | 5
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 13
Vomiting (Gastrointestinal disorders) | 2 | 5
Chills (General disorders) | 1 | 3
Edema limbs (General disorders) | 0 | 11
Edema limbs (General disorders) | 6 | 59
Fatigue (General disorders) | 3 | 27
Fever (General disorders) | 1 | 5
Gait abnormal (General disorders) | 1 | 6
General symptom (General disorders) | 1 | 1
Ill-defined disorder (General disorders) | 1 | 0
Localized edema [trunk/genital] (General disorders) | 1 | 3
Pain [NOS] (General disorders) | 1 | 1
Pain [other] (General disorders) | 3 | 10
Stern's Scale Toxicity: edema: NOS (General disorders) | 6 | 59
Gastric infection [with unknown ANC] (Infections and infestations) | 1 | 0
Infection [other] (Infections and infestations) | 0 | 4
Skin infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 1 | 1
Wound infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 2 | 10
Wound infection [with unknown ANC] (Infections and infestations) | 1 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 22
Fracture (Injury, poisoning and procedural complications) | 0 | 5
Late RT Toxicity: subcutaneous tissue: NOS (Injury, poisoning and procedural complications) | 5 | 25
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 | 10
Seroma (Injury, poisoning and procedural complications) | 1 | 10
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 5
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Alkaline phosphatase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Hyperbilirubinemia (Investigations) | 1 | 1
Laboratory test abnormal (Investigations) | 1 | 2
Leukopenia (Investigations) | 3 | 4
Lymphopenia (Investigations) | 4 | 7
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 4 | 1
Weight loss (Investigations) | 1 | 5
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatremia (Metabolism and nutrition disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint disorder (Musculoskeletal and connective tissue disorders) | 6 | 33
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 7
Late RT Toxicity: joint: NOS (Musculoskeletal and connective tissue disorders) | 6 | 30
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 5
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 40
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 4
Neuralgia (Nervous system disorders) | 2 | 4
Neurological disorder NOS (Nervous system disorders) | 0 | 4
Peripheral motor neuropathy (Nervous system disorders) | 0 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 18
Phantom pain (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Taste alteration (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 4
Depression (Psychiatric disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 4
Proteinuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 4
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Gynecomastia (Reproductive system and breast disorders) | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 | 7
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 9
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 14
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 5 | 38
Sweating (Skin and subcutaneous tissue disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 2 | 3
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 4
Vascular disorder (Vascular disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Due to unmet accrual goals for Cohort A, the decision was made to close this cohort and to increase the sample size of Cohort B. Due to the small sample size for Cohort A results were not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.